CLINICAL TRIAL: NCT03414918
Title: Macrolides for KCNJ5 - Mutated Aldosterone-Producing Adenoma (MAPA): A Study Of Personalized Diagnosis of Primary Aldosteronism With Implications For Treatment
Brief Title: Macrolides for KCNJ5 - Mutated Aldosterone-Producing Adenoma (MAPA)
Acronym: MAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Padova (Other)
Collaborators: DMG Paris Descartes (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Director of Arterial Hypertension Unit - DIMED, University Hospital Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4283/AO/17
Record Dates: First submitted 2017-12-27; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hyperaldosteronism
Keywords: Macrolides, KCNJ5 potassium channel, aldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Clarithromycin; Roxithromycin

STUDY DESIGN:
Intervention Model Description: Study 1: We will enroll consecutive hypertensive patients with PA, who need to undergo adrenal vein sampling (AVS) before being referred for adrenalectomy, according to current guidelines12.
  Study 2: Regardless of the results of study 1, we will recruit consecutive referred hypertensive patients undergoing screening for secondary hypertension. This is because to prove unambiguously the role of macrolides in the screening of mutated APA we must enroll a population of patients with and without PA and with/without the different gene mutations so far identified in APA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Clarithromycin (Experimental): 250 mg clarithromycin diluted in 250 ml saline will be administered as a slow infusion (45 min) in a peripheral vein during AVS. This dose of clarithromycin should yield peak plasma concentrations of 2.78 mcg/mL (on average)13, which are higher than the IC50 measured in vitro (0.53-1.29 mcg/mL).
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Hypertensive patients will be exposed to a single oral dose of 150 mg of roxithromycin. A 150-mg oral dose of roxithromycin should yield peak plasma concentrations of 5-12 mcg/mL14, which are higher than the IC50 measured in vitro (0.18-0.53 mcg/mL).
  Other Names: roxithromycin

SUMMARY:
This study evaluates if :

1 ) the plasma aldosterone concentration and blood pressure change in response to roxithromycin could be useful for the screening of PA patients carrying a KCNJ5-mutated APA; 2) the change of PAC in response to mutated KCNJ5 channel is truly occurring in KCNJ5-mutated APA.

DETAILED DESCRIPTION:
Aldosterone-producing adenoma (APA) cause primary aldosteronism (PA), the main curable cause of endocrine hypertension, is in up to 66% of all cases investigated with adrenal vein sampling (AVS). Mutations in the KCNJ5 potassium channel involve up to 70% of APA and cause the most florid PA phenotypes. The recent finding that macrolide antibiotics specifically inhibit in vitro the altered function of mutated KCNJ5 channels has opened new horizons for the diagnosis and treatment of APA with KCNJ5 mutations in that it can allow identification and target treatment of PA patients harbouring a mutated APA. Thus, the aim of the present study was to investigate if clarithromycin and roxithromycin, two macrolides that potently blunt mutated Kir3.4 channel function in vitro, affect plasma aldosterone concentration in adrenal vein blood during AVS and in peripheral blood, respectively, in PA patients with a mutated APA.

The investigators designed two proof of concept studies. In study A: consecutive patients with an unambiguous biochemical evidence of PA will be exposed to a single dose of 250 mg clarithromycin during AVS, to assess its effect on the relative aldosterone secretion index (RASI) in adrenal vein blood from the gland with and without APA. In study B: consecutive hypertensive patients submitted to the work-up for hypertension will receive a single oral dose of 150 mg roxithromycin. The experimental endpoints will be the change induced by roxithromycin of plasma aldosterone concentration (PAC) and other steroids, direct active renin concentration (DRC), serum K+, systolic and diastolic blood pressure.

The investigators expect to prove that: i) clarithromycin allows identification of mutated APA before adrenalectomy and sequencing of tumour DNA; ii) the acute changes of PAC, DRC, and blood pressure in peripheral venous blood after roxithromycin can be a proxy for the presence of an APA with somatic mutations.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form
* A diagnosis of hypertension defined either as:

Use of antihypertensive drug (s) Arterial hypertension: in untreated patients this must be confirmed by daytime ambulatory blood pressure monitoring (ABPM), or home blood pressure monitoring, with blood pressure higher or equal to 135 mmHg for systolic blood pressure and/or higher or equal to 85 mmHg for diastolic blood pressure.

Normal observation of ECG QT interval.

Exclusion Criteria:

* History of allergy/intolerance to any macrolides;
* Refusal of the patient to undergo dynamic testing;
* Refusal of the patient to undergo AVS and/or contraindications to the general anesthesia that is required for laparoscopic adrenalectomy (for objective 2);
* Suspicion of cortisol-aldosterone co-secreting adenoma
* Pregnancy
* Family history of sudden death
* Family history of syncope
* Family history of Long QT syndrome and or torsade de point
* Congenital or drug-induced Long QT syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Study 1: Change in Relative Aldosterone Secretion Index (RASI). | Baseline and after 45min clarithromycin infusion.
  Within-patient change from baseline of the RASI in adrenal vein blood draining the gland with and without the APA.
Study 2: Change in plasma aldosterone concentration (PAC). | Baseline and after 60 and 120 minutes roxitromycin administration
  Within-patient change from baseline of PAC in peripheral venous blood in patients undergoing screening for PA.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, MD, Principal Investigator — University of Padova
Locations (1):
- Department of Medicine - DIMED, University of Padova, Italy, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share the data will be taken upon completion of the study and publication of the results.

REFERENCES:
- [Background] Rossi GP, Belfiore A, Bernini G, Desideri G, Fabris B, Ferri C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Montemurro D, Palumbo G, Rizzoni D, Rossi E, Semplicini A, Agabiti-Rosei E, Pessina AC, Mantero F; PAPY Study Investigators. Prospective evaluation of the saline infusion test for excluding primary aldosteronism due to aldosterone-producing adenoma. J Hypertens. 2007 Jul;25(7):1433-42. doi: 10.1097/HJH.0b013e328126856e. PMID 17563566
- [Background] Choi M, Scholl UI, Yue P, Bjorklund P, Zhao B, Nelson-Williams C, Ji W, Cho Y, Patel A, Men CJ, Lolis E, Wisgerhof MV, Geller DS, Mane S, Hellman P, Westin G, Akerstrom G, Wang W, Carling T, Lifton RP. K+ channel mutations in adrenal aldosterone-producing adenomas and hereditary hypertension. Science. 2011 Feb 11;331(6018):768-72. doi: 10.1126/science.1198785. PMID 21311022
- [Background] Scholl UI, Abriola L, Zhang C, Reimer EN, Plummer M, Kazmierczak BI, Zhang J, Hoyer D, Merkel JS, Wang W, Lifton RP. Macrolides selectively inhibit mutant KCNJ5 potassium channels that cause aldosterone-producing adenoma. J Clin Invest. 2017 Jun 30;127(7):2739-2750. doi: 10.1172/JCI91733. Epub 2017 Jun 12. PMID 28604387
- [Background] Caroccia B, Prisco S, Seccia TM, Piazza M, Maiolino G, Rossi GP. Macrolides Blunt Aldosterone Biosynthesis: A Proof-of-Concept Study in KCNJ5 Mutated Adenoma Cells Ex Vivo. Hypertension. 2017 Dec;70(6):1238-1242. doi: 10.1161/HYPERTENSIONAHA.117.10226. Epub 2017 Oct 9. PMID 28993452
- [Background] Rossitto G, Battistel M, Barbiero G, Bisogni V, Maiolino G, Diego M, Seccia TM, Rossi GP. The subtyping of primary aldosteronism by adrenal vein sampling: sequential blood sampling causes factitious lateralization. J Hypertens. 2018 Feb;36(2):335-343. doi: 10.1097/HJH.0000000000001564. PMID 28957852